CLINICAL TRIAL: NCT03602560
Title: A 52-week, Placebo-controlled, Randomized, Phase 3 Study to Evaluate the Safety and Efficacy of Seladelpar in Subjects With Primary Biliary Cholangitis (PBC) and an Inadequate Response to or an Intolerance to Ursodeoxycholic Acid (UDCA)
Brief Title: ENHANCE: Seladelpar in Subjects With Primary Biliary Cholangitis (PBC) and an Inadequate Response to or an Intolerance to Ursodeoxycholic Acid (UDCA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB8025-31735
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Primary Biliary Cholangitis
Keywords: PBC; Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — seladelpar

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Seladelpar 5-10 mg (Experimental)
  Interventions: Drug: seladelpar 5-10 mg
- Seladelpar 10 mg (Experimental)
  Interventions: Drug: seladelpar 10 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: seladelpar 5-10 mg — Seladelpar 5 mg for 6 months and then titrating up to 10 mg based on tolerability and response for remainder of double-blind period. After completion of the 1-year double-blind period subjects will be offered the opportunity to enter an open label long term safety study. Subjects will continue the seladelpar dose (5 or 10 mg) received during the double-blinded study
  Arms: Seladelpar 5-10 mg
Drug: seladelpar 10 mg — Seladelpar 10 mg for double-blind period. After completion of the 1-year double-blind period subjects will be offered the opportunity to enter an open label safety study. Subjects will continue the seladelpar dose (10 mg) received during the double-blinded study
  Arms: Seladelpar 10 mg
Drug: Placebo — One capsule daily for double-blind period. After completion of the 1-year double-blind period subjects will be offered the opportunity to enter an open label long term safety study. Subjects on placebo will be re-randomized to initiate seladelpar at 5 or 10 mg once daily
  Arms: Placebo

SUMMARY:
A 52-week, placebo-controlled, randomized, Phase 3 study to evaluate the safety and efficacy of seladelpar in subjects with primary biliary cholangitis (PBC) and an inadequate response to or intolerance to ursodeoxycholic acid (UDCA)

The participants might enter the ongoing open-label safety study (NCT03301506) following this double-blind study.

DETAILED DESCRIPTION:
Primary:

* To evaluate the safety and effect on cholestasis of two seladelpar regimens (5 mg/day titrated to 10 mg/day and 10 mg/day) over 52 weeks of treatment compared to placebo

Key Secondary:

* To evaluate the effect of seladelpar on normalization of alkaline phosphatase (AP) levels
* To evaluate the effect of seladelpar on pruritus

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law
2. 18 to 75 years old (inclusive)
3. Male or female with a diagnosis of PBC, by at least two of the following criteria:

   * History of AP above ULN for at least six months
   * Positive anti-mitochondrial antibody (AMA) titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay [ELISA]) or positive PBC-specific antinuclear antibodies
   * Documented liver biopsy result consistent with PBC
4. On a stable and recommended dose of UDCA for the past twelve months OR intolerant to UDCA (last dose of UDCA > 3 months prior to Screening)
5. AP ≥ 1.67 × ULN
6. Females of reproductive potential must use at least one barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male subjects who are sexually active with female partners of reproductive potential must use barrier contraception and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose

Exclusion Criteria:

1. Previous exposure to seladelpar (MBX-8025)
2. A medical condition, other than PBC, that in the investigator's opinion would preclude full participation in the study or confound its results (e.g., cancer)
3. AST above 3 × ULN
4. ALT above 3 × ULN
5. Total bilirubin above 2.0 × ULN
6. Advanced PBC as defined by the Rotterdam criteria (albumin below LLN AND total bilirubin above 1 × ULN)
7. Creatine kinase (CK) above 1.0 × ULN
8. eGFR below 60 mL/min/1.73 m2 (calculated by MDRD formula)
9. International normalized ratio (INR) above 1.0 × ULN
10. Platelet count below 100 × 103/µL
11. Presence of clinically significant hepatic decompensation, including:

    * History of liver transplantation, current placement on liver transplantation list, or current MELD score ≥ 15
    * Complications of portal hypertension, including known esophageal varices, history of variceal bleeds or related interventions (e.g., transjugular intrahepatic portosystemic shunt placement), relevant ascites, hepatic encephalopathy
    * Cirrhosis with complications, including history or presence of spontaneous bacterial peritonitis
12. Other chronic liver diseases:

    * Current features of auto-immune hepatitis as determined by the investigator based on immunoserology, liver biochemistry and histology
    * Primary sclerosing cholangitis determined by presence of diagnostic cholangiographic findings
    * History or clinical evidence of alcoholic liver disease
    * History or clinical evidence of alpha-1-antitrypsin deficiency
    * Biopsy confirmed nonalcoholic steatohepatitis
    * History or evidence of Gilbert' Syndrome with elevated total bilirubin
    * History or evidence of hemochromatosis
    * Hepatitis B defined as presence of hepatitis B surface antigen (HBsAg)
    * Hepatitis C defined as presence of HCV RNA
13. Known history of HIV
14. Evidence of significant alcohol consumption
15. Evidence of drug abuse
16. Subjects with inadequate response to obeticholic acid (OCA) or intolerance to OCA: OCA must be discontinued 30 days prior to Screening
17. Use of colchicine, methotrexate, azathioprine, or long-term systemic corticosteroids (> 2 weeks) within two months prior to Screening
18. Use of fibrates within 30 days prior to Screening
19. Use of simvastatin within 7 days prior to Screening
20. Use of an experimental or unapproved treatment for PBC within 30 days prior to Screening
21. Use of experimental or unapproved immunosuppressant within 30 days prior to Screening
22. Treatment with any other investigational therapy or device within 30 days or within five half-lives, whatever is longer, prior to Screening
23. For females, pregnancy or breast-feeding
24. Any other condition(s) that would compromise the safety of the subject or compromise the quality of the clinical study, as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (156):
- United States (51):
  - Institute for Liver Health, Chandler, Arizona
  - Mayo Clinic Arizona - PPDS, Phoenix, Arizona
  - The Institute for Liver Health-Tucson, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Redwood City, California
  - University of California Davis Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Univeristy of Colorado Denver and Hospital, Aurora, Colorado
  - Yale School of Medicine Digestive Diseases, Internal Medicine, New Haven, Connecticut
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Florida Reserach Institute, Lakewood Rch, Florida
  - Schiff Center for Liver Diseases University of Miami, Miami, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Minnesota Gastroenterlogy, P.A., Maplewood, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Southern Therapy and Advance Research (STAR) LLC, Jackson, Mississippi
  - Digestive Health Specialists PA, Tupelo, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Concorde Medical Group, New York, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Center for Liver Disease and Transplantation, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Asheville Gastroenterology Associates, a Division of Digestive Health Partners, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - GIA Clinical Trials, LLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Liver Institute at Methodist Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Digestive Disease Consultants, Fort Worth, Texas
  - American Research Corporation, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Mary Immaculate Hospital, Newport News, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- Argentina (4):
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Fundación Sanatorio Güemes, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital Provincial Del Centenario, Rosario, Santa Fe Province
  - DIM Clínica Privada, Ramos Mejía
- Australia (5):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (4):
  - Medizinische Universitat Wien, Vienna, Vienna
  - LKH-Universitätsklinikum Klinikum Graz, Graz
  - Salzburger Landeskliniken, Salzburg
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
- Canada (5):
  - University of Calgary Medicine, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - University Health Network, Toronto, Ontario
  - Toronto Digestive Disease Associates Inc, Vaughan, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- Chile (3):
  - Pontificia Universidad Catolica de Chile, Santiago, Región-MetropolitanadeSantiago
  - Centro Clinico Mediterraneo, La Serena
  - Centro de Investigaciones Clínicas Vina del Mar, Viña del Mar
- France (3):
  - Hôpital Jean Verdier, Bondy
  - CHU de GRENOBLE, Grenoble
  - Hôpital Saint Antoine, Paris
- Germany (8):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne, North Rhine-Westphalia
  - Gastroenterologisch Hepatologisches Zentrum Kiel, Kiel, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - ifi-Institute for Interdisciplinary Medicine, Hamburg
  - Universitatsklinikum Leipzig, Leipzig
- Greece (3):
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
- Hungary (4):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Budai Hepatológiai Centrum, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- Israel (8):
  - Hillel Yaffe Medical Center, Hadera
  - Carmel Medical Center, Haifa
  - Rambam Health Corporation, Haifa
  - Hadassah Medical Center, Jerusalem
  - The Galilli Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - ASST Santi Paolo e Carlo - Azienda Universitaria-Polo Universitario San Paolo, Milan
  - Ospedale Civile di Baggiovara, Modena
  - Azienda Ospedaliera Di Padova, Padua
  - ASST di Monza - Azienda Ospedaliera San Gerardo, Rozzano
- Mexico (3):
  - Centro de Diabetes y Obesidad Graber, Pachuca, Hidalgo
  - Consultorio de la Doctora Maria Sarai Gonzalez Huezo, Metepec
  - Consultorio Medico - Distrito Federal, Mexico City
- Radboud Universitair Medisch Centrum, Nijmegen, Gelderland, Netherlands
- New Zealand (3):
  - Christchurch Hospital, Christchurch, South Island
  - Dunedin Hospital, Dunedin, South Island
  - Waikato Hospital, Hamilton
- Poland (6):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 7 Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice, Silesian Voivodeship
  - Wojewodzki Szpital Zespolony w Kielcach, Kielce
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - ID Clinic, Mysłowice
- Romania (4):
  - Pius Brinzeu Emergency Clinical County Hospital, Timișoara, Timiș County
  - Colentina Clinical Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Sana Monitoring SRL, Bucharest
- Russia (3):
  - Peoples Friendship University of Russia, Moscow, Moscow
  - City Hospital #31, Saint Petersburg
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
- Serbia (2):
  - Clinical Hospital Centar Zvezdara, Belgrade
  - KBC Zemun, Belgrade
- South Korea (8):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Inje University Ilsan Paik Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (10):
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (10):
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - University Hospital Birmingham, Birmingham
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Barts Health NHS Trust, Royal London Hospital, Ambrose King Centre, London
  - Royal Free London NHS Foundation Trust, London
  - Kings College Hospital, London
  - The Newcastle Upon Tyne Hospital NHS Foundation Trust, Newcastle
  - University of Nottingham, Nottingham
  - Plymouth Hospitals NHS Trust, Plymouth
  - Singleton Hospital, Swansea

RESULTS

PARTICIPANT FLOW:
Groups:
- Seladelpar 5-10 mg: seladelpar 5-10 mg: Seladelpar 5 mg for 6 months and then titrating up to 10 mg based on tolerability and response for remainder of double-blind period.
- Seladelpar 10 mg: seladelpar 10 mg: Seladelpar 10 mg for double-blind period.
- Placebo: Placebo: One capsule daily for double-blind period.
Period: Overall Study
Arm/Group | Seladelpar 5-10 mg | Seladelpar 10 mg | Placebo
Started | 89 | 89 | 87
Completed | 1 | 1 | 1
Not Completed | 88 | 88 | 86

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seladelpar 5-10 mg | Seladelpar 10 mg | Placebo | Total
Number analyzed (Participants) | 89 | 89 | 87 | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 73 | 73 | 221
  >=65 years | 14 | 16 | 14 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 83 | 85 | 250
  Male | 7 | 6 | 2 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 4 | 8 | 5 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 2 | 7
  White | 83 | 77 | 80 | 240
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response to Composite Endpoint of ALP <1.67 × Upper Limit of Normal [ULN], ≥15% Reduction in ALP, and Total Bilirubin ≤ ULN) at Month 3
Description: Percentage of Participants with Response to Composite Endpoint of ALP <1.67 × Upper Limit of Normal [ULN], ≥15% reduction in ALP, and total bilirubin ≤ ULN) at Month 3. The mITT analysis set included all randomized subjects who received at least one study drug dose.
  The primary endpoint was analyzed using Cochran-Mantel-Haenszel (CMH) test adjusted for both randomization stratification variables (ALP level: <350 U/L and 2:350 U/L; pruritus NRS: <4 and 2:4). The CMH tests were performed for the comparison of 10 mg versus placebo and 5 mg/10 mg versus placebo separately.
Time Frame: Month 3
Population: mITT Population. The Modified Intent-to-Treat (mITT) set includes any subject who is randomized into the study and receives at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 5-10 mg | Seladelpar 10 mg | Placebo
Number analyzed (Participants) | 56 | 55 | 56
Participants | 32 | 43 | 7
Statistical Analysis 1: Comparison: Seladelpar 10 mg vs Placebo; Test type: Other — The primary endpoint was analyzed using Cochran-Mantel-Haenszel (CMH) test adjusted for both randomization stratification variables (ALP level: <350 U/L and 2:350 U/L; pruritus NRS: <4 and 2:4); p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Seladelpar 5-10 mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With Response Defined by Normalized Alkaline Phosphatase Levels at Month 3
Description: The response was defined by normalized ALP levels (ALP ≤1.0 × ULN) at endpoint. The mITT analysis set included all randomized subjects who received at least one study drug dose.
Time Frame: Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Seladelpar 5-10 mg | Seladelpar 10 mg | Placebo
Number analyzed (Participants) | 56 | 55 | 56
Participants | 3 | 15 | 0
Statistical Analysis 1: Comparison: Seladelpar 10 mg vs Placebo; Test type: Other — Two-sided p-value for each pair-wise comparison was based on the CMH test adjusted for both randomization stratification variables (ALP level: <350 U/L and 350 U/L; pruritus NRS: <4 and 4). Breslow-Day test was used to check the homogeneity of treatment effects across stratum; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Seladelpar 5-10 mg vs Placebo; Test type: Other — Two-sided p-value for each pair-wise comparison is based on the Cochran Mantel Haenszel test adjusted for both randomization stratification variables (ALP level: < 350 U/L and >= 350 U/L; pruritus NRS: < 4 and >= 4). Breslow-Day test is used to check the homogeneity of treatment effects across stratum; p = 0.0839, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in Pruritus NRS for Subjects With Baseline NRS ≥4 at Month 3
Description: Pruritus Numerical Rating Scale (NRS) used to rate the intensity of the worst itching you experienced in the past 24 hours from no itching to worst possible itching by selecting a number from 0 to 10 on Itch Scale. Zero means no itching and 10 means worst imaginable itching. The analysis will be limited to those subjects in the mITT analysis set with a baseline NRS ≥ 4.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seladelpar 5-10 mg | Seladelpar 10 mg | Placebo
Number analyzed (Participants) | 17 | 18 | 18
score on a scale | -1.95 (2.226) | -3.01 (1.952) | -1.44 (1.831)
Statistical Analysis 1: Comparison: Seladelpar 10 mg vs Placebo; Test type: Other — Change from baseline is estimated by an analysis of covariance (ANCOVA) model with treatment group (including 3 levels: Placebo, Initial Dose 5mg, and Initial Dose 10 mg) and randomization ALP stratification as factors, and baseline as a covariate. The p-value for the interaction between treatment and stratum is 0.7595, hence the interaction is dropped from the model; p = 0.0164, ANCOVA; Risk Difference (RD) = -1.59, 95% CI 2-sided [-2.87 to -0.3]
Statistical Analysis 2: Comparison: Seladelpar 5-10 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.4781, ANCOVA; Risk Difference (RD) = -0.46, 95% CI 2-sided [-1.77 to 0.84]

ADVERSE EVENTS:
Time Frame: An AE will be recorded any time after the time of signed ICF and captured until this double-blinded study's last study visit, up to 1 year.
Groups:
- Seladelpar 5/10 mg: Seladelpar 5/10 mg in this double-blinded study
- Seladelpar 10 mg: Seladelpar 10 mg in this double-blinded study
- Placebo: Placebo in this double-blinded study
Arm/Group | Seladelpar 5/10 mg | Seladelpar 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/89 | 0/87
Serious Adverse Events (participants affected / at risk) | 3/89 | 1/89 | 3/87
Other Adverse Events (participants affected / at risk) | 55/89 | 58/89 | 62/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seladelpar 5/10 mg (N=89) | Seladelpar 10 mg (N=89) | Placebo (N=87)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seladelpar 5/10 mg (N=89) | Seladelpar 10 mg (N=89) | Placebo (N=87)
Dry eye (Eye disorders) | 3 (3) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 6 (6) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (6) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 7 (8) | 4 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Asthenia (General disorders) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (4) | 8 (8)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 7 (8) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 10 (11) | 11 (16)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03602560/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT03602560/SAP_001.pdf